CLINICAL TRIAL: NCT00476164
Title: Randomised Trial of Anti-Cd20 in C4d+ Chronic Allograft Nephropathy
Brief Title: Study of Rituximab to Treat Chronic Renal Transplant Rejection
Acronym: RituxiCAN-C4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Medical Research Council (Other Government); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, A. Dorling, Professor of Transplant Inflammation and Repair, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-002330-38
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Kidney Transplantation; Graft Rejection; Immunosuppression
Keywords: chronic allograft nephropathy; C4d; Anti-CD20; B cells; Antibody
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Infusion of 2 x 1g of rituximab, 14 days apart
  Interventions: Drug: Rituximab
- 2 (Sham Comparator)
  Interventions: Other: Control arm

INTERVENTIONS:
Drug: Rituximab — 2 doses of 1g 14 days apart
  Other Names: Mabthera
  Arms: Rituximab
Other: Control arm — Continue of optimised oral immunosuppression
  Arms: 2

SUMMARY:
Purpose of clinical trial; Evaluate the effectiveness of rituximab in C4d+ CAN

Primary objective; To determine whether anti-CD20 therapy can stabilize or improve renal function and/or proteinuria in patients with C4d+, chronic (humoral) rejection in whom standard therapeutic approaches have failed.

Secondary objective (s);

* To compare patient and graft survival between control and rituximab-treated groups
* To evaluate the adverse effect profile of rituximab in this group
* To correlate changes in circulating B cell numbers, anti-HLA and non-HLA Ab profiles and titre with responses to standard therapy and / or rituximab
* To correlate changes in T cell responsiveness to alloantigens with responses to standard therapy and / or rituximab

Study Design; Prospective, randomised, two arm, open-labeled

Study Endpoints; Primary

* Rate of deterioration in renal function, defined by slope of reciprocal creatinine plot, on samples taken 3-5 months post-randomisation.
* Change in degree of proteinuria, where present, at 3-5 months post-randomisation 2˚ endpoints, determined at 3-5 months post-randomisation and at 1, 2 and 3 years post-recruitment are;
* Rate of deterioration in renal function, defined by slope of reciprocal creatinine plot, determined by analysis of samples taken since previous assessment.
* Patient survival
* Graft survival
* Incidence of culture positive infection
* Incidence of malignancy
* Degree of proteinuria
* Changes in circulating CD20+ cells in peripheral blood
* Changes in anti-graft Ab titres, (measured every 3 months)
* Changes in T cell responsiveness to alloantigens (measured every 3 months).

Sample Size; 15 patients to be randomised to each arm (i.e. 30 patients randomised). Up to 120 patients will need to be enrolled into the study. In addition, in those participants that received a living donor kidney, these donors will be approached to provide up to 5 samples of blood to help with the in vitro analyses.

Summary of eligibility criteria;

* Male or female renal allograft recipients 18-70 years of age
* more than 6/12 post-transplantation
* Either deteriorating allograft function on reciprocal creatinine plot or significant proteinuria or both.
* C4d+/- CAN on renal allograft biopsy

Investigational medicinal product and dosage; Rituximab, 1g on day 0 and 1g on day 14

Active comparator product(s); None

Route(s) of administration; Intravenous infusion

Maximum duration of treatment of a subject; 14 days with rituximab. The treatment arms of the study, including optimisation period, formal run-in and post-randomisation phase lasts for 10 months post-recruitment.

Procedures; Screening & enrollment. Potentially eligible patients will be identified by screening renal allograft biopsies performed for 'creeping creatinine' and/or proteinuria. Recruitment by informed consent prior to enrollment.

Procedures; Baseline. In addition to routine tests, blood for anti-HLA and non-HLA antibody analysis and for peripheral blood mononuclear cell (PBMC) purification.

Procedures; Treatment period. 3 month run-in period on optimal conventional immunosuppressive therapy, preceded by up to 2 months to allow tailored-optimization. Patients will be reviewed at least six times in their normal transplant clinic appointments for routine blood biochemistry, full blood count and urine analysis. At the end of the run-in period, further blood will be taken for anti-graft antibody analysis and PBMC purification. Those patients in whom allograft function stabilises and/or proteinuria improves will have normal transplant clinic follow-up appointments and have blood taken for further anti-graft antibody and PBMC purification up to every 3 months for 3 years. Those with continued deterioration in either allograft function or persisting or worsening proteinuria will be randomised. These patients will be reviewed during their normal transplant clinic appointments until the primary end-point and will need to have at least 6 routine blood biochemistry, full blood count and urine analysis during the final 3 months of this period, post-randomisation. At the primary end-point, further blood will be taken for anti-graft antibody analysis and PBMC.

Procedures; End of Study. •Follow up will continue for 3 years, with blood taken for anti-graft antibody analysis and PBMC purification every three months

Procedures for safety monitoring during trial; Regular patient interviews and examination, routine haematological and biochemical analyses. Serious adverse events will be reported and forwarded to the sponsor, MHRA, LREC and Roche as appropriate The WLRATC transplant research committee will discuss the trial and any safety concerns at their regular three monthly meetings. Data will be reviewed after 30 and also after 60 people have been enrolled.

Criteria for withdrawal of patients on safety grounds; Serious adverse effects related to rituximab infusion

ELIGIBILITY:
Inclusion Criteria:

* Functioning kidney allograft (with estimated (e) GFR by MDRD >20) and be >6/12 post-transplantation
* Deteriorating allograft function as defined by linear regression of reciprocal creatinine plot. Deterioration will be defined as a negative slope over at least the preceding 3 months (with at least 6 creatinines included) with an adjusted r2 >0.35 and a p value of ≤0.05 compared to horizontal baseline. Deterioration will be confirmed by reduction in Cockcroft-Gault (CG) eGFR over the same period (to exclude increases in body mass as a cause of a negative slope on reciprocal creatinine plots) OR significant proteinuria as assessed by a urine protein/creatinine ratio of ≥50
* CAN, by Banff '97 criteria, and/or transplant glomerulopathy on renal allograft biopsy performed within 6/12 of enrolment
* Diffuse, linear C4d deposition on at least 25% of peritubular capillary (PTC) and/or glomerular EC of renal transplant biopsy when assessed by immunoperoxidase or >50% of PTC (alone) when assessed by immunofluorescence OR PTCitis OR glomerulitis with combined PTC/g score of ≥2.

Exclusion Criteria:

* Ages below 18 years of age
* Suspicion of pregnancy confirmed by positive HCG pregnancy test
* Untreated ureteric obstruction on ultrasound of allograft
* History of acute allograft rejection in preceding 3/12
* History of MI in preceding 3/12
* History of malignancy in previous 5 years (excluding tumours limited to skin)
* Symptomatic IHD
* Recipient of simultaneous pancreas/kidney transplant
* Recipient of ABO-incompatible kidney
* Recipient who underwent an HLA desensitisation procedure prior to transplantation
* Evidence, on examination of renal allograft biopsy specimen, of recurrent or de-novo disease (except IgA deposition in absence of mesangial proliferation)
* Evidence, on examination of renal allograft biopsy specimen, of CNI toxicity IF ACCOMPANIED by mostly supra-therapeutic CNI trough levels in the 6 month period preceding biopsy.
* Documented allergy to mouse or chimeric human/mouse proteins
* HepBsAg+, HepBcAb+, HCV Ab+ or HIV+.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-01; Primary Completion 2015-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Rate of deterioration in renal function, defined by slope of reciprocal creatinine plot | 3-5 months post-randomisation
Change in degree of proteinuria, where present | 3-5 months post-randomisation

SECONDARY OUTCOMES:
Rate of deterioration in renal function, defined by slope of reciprocal creatinine plot, determined by analysis of samples taken since previous assessment | 1, 2 and 3 years post-recruitment
Patient survival | 5 months post-randomisation and at 1, 2 and 3 years post-recruitment
Graft survival | 5 months post-randomisation and at 1, 2 and 3 years post-recruitment
Incidence of culture positive infection | 5 months post-randomisation and at 1, 2 and 3 years post-recruitment
Incidence of malignancy | 5 months post-randomisation and at 1, 2 and 3 years post-recruitment
Degree of proteinuria | 1, 2 and 3 years post-recruitment
Changes in circulating CD20+ cells in peripheral blood | 5 months post-randomisation and at 1, 2 and 3 years post-recruitment
Changes in anti-graft Ab titres | 3 monthly to 3 years post-recruitment
Changes in T cell responsiveness to alloantigens | 3 monthly to 3 years post-recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Dorling, PhD FRCP, Principal Investigator — King's College London
Locations (11):
- United Kingdom (11):
  - University Hospital Birmingham, Birmingham
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Univeristy Hospital of Wales, Cardiff
  - Epsom & St Helier University Hospitals Trust, Carshalton
  - Western Infirmary, Glasgow
  - Hull Royal Infirmary, Hull
  - St Jame's University Hospital, Leeds
  - The Royal Free Hospital, London
  - King's College London, Guy's Hospital, London
  - Imperial College London and West London Renal & Transplantation Centre, London
  - Manchester Royal Infirmary, Manchester

REFERENCES:
- [Result] Shiu KY, Stringer D, McLaughlin L, Shaw O, Brookes P, Burton H, Wilkinson H, Douthwaite H, Tsui TL, Mclean A, Hilton R, Griffin S, Geddes C, Ball S, Baker R, Roufosse C, Horsfield C, Dorling A. Effect of Optimized Immunosuppression (Including Rituximab) on Anti-Donor Alloresponses in Patients With Chronically Rejecting Renal Allografts. Front Immunol. 2020 Feb 5;11:79. doi: 10.3389/fimmu.2020.00079. eCollection 2020. PMID 32117242
- See also: Pre-print version of the manuscript describing the trial outcomes — https://kclpure.kcl.ac.uk/portal/en/publications/effect-of-optimised-immunosuppression-including-rituximab-on-antidonor-alloresponses-in-patients-with-chronically-rejecting-renal-allografts(701fe5d0-440a-49fb-9ab2-28dfcccca876).html
- See also: Full print version of trial outcomes manuscript — https://www.frontiersin.org/articles/10.3389/fimmu.2020.00079/full